Fluoxetine to Reduce the Risk of Morbidity and Mortality with COVID-19 Infection Cheryl McCullumsmith, MD PhD, Principal Investigator NCT04377308 May 2, 2020

# Fluoxetine to reduce the risk of morbidity and mortality with COVID-19 infection

Cheryl McCullumsmith, MD PhD, Principal Investigator

# 1. Background, Review of the Literature, Significance

Much of the morbidity and mortality with COVID-19 infection is thought to be the result of multisystem organ failure after a cytokine storm (Huang et al. *Lancet* 2020). This cytokine storm is very similar if not identical to the Secondary Hemophagochytic Lymphohistiocytosis (SHLH) seen in Severe Acute Respiratory Syndrom (SARS) also caused by a coronavirus, and includes increased levels of IL-2, IL-7, C-CSF, TNF-2, interferon-G inducible protein, MCP1 and MIP1a, all of which are driven by increased levels of IL-6. (Taraz 2013, Gobin, 2014) These findings have led to use of medications such as tocilizumab, an IL-6 receptor antagonist, to treat COVID-19 pneumonia. Fluoxetine and certain other selective serotonin reuptake inhibitors (SSRIs) have demonstrated in vitro and in vivo efficacy at reducing IL-6 and both preventing and treating hyperimmune responses associated with elevated levels of IL-6. Further, fluoxetine has a very safe therapeutic profile and could be used both prophylactically to prevent the cytokine storm with COVID-19, as well as an adjuvant treatment for critically ill patients.

*In vitro* and *in vivo* data demonstrate that fluoxetine and some other selective serotonin reuptake inhibitors (SSRIs) effectively reduce IL-6 to prevent hyperimmune response. In addition to SSRI use in adjuvant treatment for critically ill patients, the established safety profiles of many SSRIs allow these drugs to be used prophylactically in order to prevent cytokine storm associated with COVID-19 infections. SSRI treatment before starting antiviral therapies reduces incidence of interferon-induced depression and carries minimal side effect profiles consisting of rare dizziness (Udina et al., 2014). The SSRI fluoxetine demonstrates a particularly pronounced ability to inhibit IL-6 activation (Durairaj, Steury, & Parameswaran, 2015; Hashioka et al., 2007). This effect is mediated by non-serotonergic pathways involving NF-kB suppression and inhibition of dendritic cell antigen presentation (Branco-de-Almeida et al., 2011; D. Liu et al., 2011; R. P. Liu et al., 2014; Vollmar, Haghikia, Dermietzel, & Faustmann, 2008; Young et al., 2014). Animal models demonstrate that SSRIs protect against hyperinflammatory conditions and diseases states. In fact, pretreatment with fluoxetine frequently outperforms pretreatment with corticosteroids (Dong et al., 2016). Recently, clinical trials have demonstrated compelling relationships between SSRI treatment and cytokine levels (Amitai et al., 2016). A recent 2019 review and meta-analysis by Wang et al. echoes previous animal work and suggests that SSRI therapy indeed reduces IL-6 levels in human subjects (Wang et al., 2019).

These data are significant to COVID-19 patients at risk for pulmonary symptoms. Pretreatment with SSRIs results in decreased destructive immune reactions across a variety of animal models. In rat models of chronic obstructive pulmonary disease, fluoxetine decreases lung injury and inhibits cytokines such as TNF-a and IL-6 (Cai et al., 2017). Indeed, fluoxetine reduces inflammatory reaction in several models of human disease, providing marked decreases in reactive cytokines (Roumestan et al., 2007). In addition to decreasing expression of inflammatory cytokines, pretreatment with fluoxetine also decreases incidence of pulmonary arterial hypertension, pulmonary arterial muscularization, and extracellular matrix remodeling (Li et al., 2011). Bronchial asthma models show therapeutic effects of fluoxetine pretreatments in rats (Sherkawy, Abo-Youssef, Salama, & Ismaiel, 2018), and several studies suggest positive therapeutic efficacy may be concurrent with reduced levels of cytokines including IL-6 (Blatteau et al., 2012; Blatteau et al., 2015).

Overall, there is significant preclinical data supporting the use of SSRI's in the abrogation of harmful inflammatory side effects, such as those driving COVID19 morbidity and mortality. Furthermore, clinical data shows robust safety and efficacy profiles supporting the use of fluoxetine pretreatment interventions. At the University of Toledo Medical Campus, we are fortunate to have a leading expert on the relationship between antidepressant drugs and their anti-inflammatory therapeutic effects. Dr. Kevin Pan, who will be leading the laboratory work described in this proposal, has published extensively on the use of antidepressants to limit organ damage, decrease pro-inflammatory cytokine production, and inhibit intracellular migration of early-stage inflammatory response (Lu, Wang, Chen, Jiang, & Pan, 2020). A recent Nature publication from Dr. Pan and his team explore connections between antidepressant drug administration and cytokine signaling, providing compelling support for the use of antidepressants in inflammatory disease states. Several studies from Pan et al. indicate antidepressant use inhibits pro-inflammatory cytokine gene expression both *in vitro* and *in vivo*. Using Dr. Pan's methods, we will assay and investigate cytokine expression in our control and experimental patients while utilizing the expertise that Dr. Pan and his University of Toledo researcher team has developed on this topic.

Further evidence for the efficacy of fluoxetine in decreasing the IL-6 response that stimulates the cytokine storm in COVID-19 infection comes from an analysis comparing the transcriptomes of cells lines treated with fluoxetine, dexamethasone (a steroid established to decrease IL-6), and 2 other antidepressants: bupropion and paroxetine to the transcriptome of the same cell line with a knock down in the IL-6 signal transduction molecule. This analysis was performed this week in the bioinformatics group in the Department of Neurosciences at University of Toledo and is illustrated

below. The concordance of the fluoxetine and IL-6ST knockdown cell lines is remarkably high, averaging over 0.7. This concordance is greater than that seen with dexamethasone treatment, the standard anti-inflammatory steroid, and is higher than 2 other commonly used antidepressants, bupropion and paroxetine.



# 2. Objectives/Specific Aims

**Aim 1:** Fluoxetine treatment begun early after COVID-19 infection will reduce hospitalizations, intubations, and death from COVID-19 and complications more than no medication

**Aim 2:** Fluoxetine will decrease intubations and mortality in patients hospitalized with COVID-19 infection greater than no medication.

**Aim 3**: Fluoxetine treatment of COVID-19 infected patients will not cause significant side effects or increase morbidity and mortality compared to no medication

**Aim 4.** Collect blood samples from 40 subjects for future cytokine analysis: both subjects taking fluoxetine and not taking fluoxetine samples taken at baseline and weekly after study initiation.

#### 3. Methods

a) Study Design: Pragmatic Clinical Trial: Experimental and Observational

# b) Method of treatment assignment

Single arm patient centered clinical trial

At study entry, participants will consent study participation via daily monitoring and will choose whether to participate in the activity monitoring, cytokine assessment and drug treatment portions of the trial. Participants who do not choose to take fluoxetine will serve as the control subjects. Additionally, patients will have the choice weekly to decide to start, continue, or discontinue the fluoxetine. See figure below:



#### c) Inclusion/exclusion criteria

Inclusion: Patients aged 18 and above, able to give informed consent

COVID-19 test positive or presumptive positive awaiting COVID testin or results by following criteria: fever, cough and shortness of breath

# Overall Study Exclusion Criteria:

Unable to give informed consent

Prisoner/ institutionalized patient

Under age 18

#### Exclusion from Fluoxetine Arm:

Active bleeding requiring blood products

Bipolar disorder not on mood stabilizing medication\*

Known allergy or hypersensitivity to fluoxetine

Currently taking the following medications: MAO I, pimozide, thioridine

Currently taking hydroxychloroquine

Pregnant or breastfeeding (pregnancy questionnaire attached)

For hospitalized patients: QTc greater than 500 ms

\*Hospitalized patient may be on hydroxychloroquine if QTc<500 and the primary attending approves

### Exclusion from Blood Sample Provision:

Pregnant

Self-report of under 110 pounds

## d) Justification of the number of subjects

All power calculations were done with the clincalc program and assume a dichotomous endpoint in a two independent sample study and are based on achieving the standards of a power of 0.80 and with an alpha of 0.05. Please note, that the assumptions of fluoxetine effect size are based on the absolute most conservative values in the published literature reviewed above.

#### Aim 1: Hospitalization rates

#### Assumptions:

- 1. 2/3 of patients who enter the trial will choose to take fluoxetine
- 2. 10% of COVID-19 + patients will progress to a clinical condition requiring hospitalization
- 3. Fluoxetine treatment decreases hospitalization rate by 50%

Sample Size: 312 in the no medication group and 624 in the 2 fluoxetine groups, for a total sample size of 936. This sample size is very achievable given the current coronavirus pandemic.

# **Prevention of Hospitalization**

| Total | 936 |
|--------------------------------|------|
| Fluoxetine, low or high | 624 |
| No medication | 312 |
| Sample Size | |
| Power | 0.8 |
| Beta | 0.2 |
| Alpha | 0.05 |
| Hospitalization, Fluoxetine | 5% |
| Hospitalization, no medication | 10% |

Aim 2: Intubation in those hospitalized

# Assumptions

- 1. 10% of patients requiring hospitalization for COVID-19 + will progress to intubation
- 2. Fluoxetine treatment decreases intubation rate by 20%

# Aim 2: Death in those hospitalized

#### Assumptions

- 1. 1% of patients requiring hospitalization for COVID-19 + will die during that hospitalization
- 2. Fluoxetine treatment decreases mortality rate by 20%

**Sample Size**: 3213 in the no medication group and 3213 in the fluoxetine groups, for a total sample size of 6426. These sample sizes will not be achievable in this pilot study. Data from Aims 3 and 4 will therefore be used qualitatively for the gathering of pilot data.

| Prevention of intubation, death | |
|---------------------------------|------|
| Sample Size | |
| No medication | 3213 |
| Fluoxetine | 3213 |
| Total | 6426 |
| Prevention of Intubation | |

| Intubation, death in no medication | 10% |
|------------------------------------|------|
| Intubation, death in fluoxetine | 8% |
| Alpha | 0.05 |
| Beta | 0.2 |
| Power | 0.8 |

# e) Study setting

Telephone, outpatient offices, emergency department, Hospital

# f) Primary and secondary outcome measures

# **Primary Outcome Measures:**

Aim 1: Rates of Hospitalization

Aim 2: Rates of Intubation and Death

Aim 3 : Side effect profile

**Secondary Outcome Measures:** 

Aim 1 and 2: Depression, Anxiety, Suicidal thinking, Days of Illness, Severity of Illness

## g) Variables

| Demographic information (age, gender, medical history, co-morbidities, etc.) |
|------------------------------------------------------------------------------|
| Medications |
| Symptom profile |
| Number of days of symptoms prior to testing |
| Epidemiologic information from CDC/Health Department surveillance interview |
| Hospital Course |
| Days in Hospital, Intubation, Complications |
| Outcome: Never hospitalized, Hospitalized, Intubation, Death |

# h) Procedures, interventions, schedule

| Week/Day | Day Patient Intervention Setting/ | | Standard | Research |
|---|---|---|---|---|
| | | Responsible | of Care | <b>Purposes Only</b> |
| | | Individual | | |
| 1/1 | Informed Consent | Phone/ research team | | Yes |
| 1/1 | Baseline Study Data | Phone/ research team | | Yes |
| 1 | Blood Sample | Laboratory Services | Inpatient | outpatient |
| 1 | Physician Interview/ | Phone/Study | | Yes |
| | Medication Prescription | physician | | 1 CS |
| Daily | Symptom/ Side effect | Phone/ research team | | Yes |
| | Check In | | | 1 05 |
| Weekly | Physician Interview/ | Phone/Study | | Yes |
| Medication Prescription physi | | physician | | 1 CS |
| Weekly or | Blood Sample | Laboratory Services | | |
| Change in | | | Inpatient | outpatient |
| Clinical | | | inpatient | Outpatient |
| Status* | | | | |

<sup>\*</sup>Change in Clinical Status includes outpatient to inpatient, transfer to ICU, and intubation

# **Procedures**:

| Instrument | Duration | Assessment Time<br>Points | Frequency |
|---|---|---|---|
| Baseline Intake Form | 30 min | Initial study entry | Once |
| Chart Review Form | | | |
| 04/1/19-present | | | |
| Baseline Demographics and past | | | |
| medical history | | | |
| PHQ-9 | 5 min | Initial Study Entry | Weekly |
| GAD-7 | 5 min | Initial Study Entry | Weekly |
| Columbia Screener-recent | 3 min | Initial study Entry | |
| Symptom Checklist | 5 min | (included in baseline) | Daily assessments |
| Columbia Screener – since last | 3 min | | Daily assessments |
| visit | | | - |
| Physician Interview/Medication | 40 min | Baseline | weekly |
| Prescription | | | - |

| Drug Distribution | | Once, at entry | monthly |
|---|---|---|---|
| Blood Draw for future | 60 min | Baseline | Weekly, as possible |
| assessment of cytokine levels | | | |
| Chart Review Followup | | At study exit, one month, 3 months, 6 months and one year after study exit | See notes to left<br>5 data points<br>From 4/1/19- 4/1/23 |

## Physician Interview/Medication Prescription

#### Interview includes:

- 1) Assessment for pregnancy, contraindicated medications and review of baseline intake
- 2) Explanation of risks and benefits of medication : see patient handout information sheet Blood Draw for Future Assessment of Cytokine Levels :
  - Not to exceed 2 blood draws per week or a total of 50 ml total over 8 weeks time period
  - Outpatient blood draws will occur only if study participants have regular clinical care blood
    draws until adequate personal protection equipment (PPE) is available for use in research
    settings. Study outpatient blood draw will occur by appointment at UTMC Emergency
    Department in a negative pressure room. Outpatient blood draws will not be done until there is
    adequate PPE available for research study purposes.
    - o Study participant and phlebotomist will be equipped in full PPE.
  - Inpatient blood draws will occur during normal clinical care blood draws.
  - Blood samples will be stored at -80 degrees F in the hospital laboratory freezers for future cytokine analysis

# **Study Timeline:**

Fluoxetine to reduce the risk of morbidity and mortality with COVID-19 infection

| 10 | ID Task Name Start Finish Duration | Tarli Nama | rinink | 5.11 | Q2 20 | | | Q3 20 | | | Q4 20 | | | Q1 21 | | | Q2 2 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | | Apr | May | Jun | Jul | Aug | Sep | Oct | Nov | Dec | Jan | Feb | Mar | Apr | May | Jun | |
| 1 | Enroll Patients in Overall Study | 4/1/2020 | 4/1/2021 | 262d | | | | | | | | | | | | | |
| 2 | Enroll Patients in Fluoxetine Arm | 4/1/2020 | 2/1/2021 | 219d | | | | | | | | | | | | | |
| 3 | Enroll Patients in Cytokine Study | 4/1/2020 | 10/1/2020 | 132d | | | | | | | | | | | | | |
| 4 | Data Analysis | 7/1/2020 | 7/1/2021 | 262d | | | | | | | | | | | | | |
| 5 | DSMB Review 1 | 7/1/2020 | 7/1/2020 | 1d | | | | 1 | | | | | | | | | |
| 6 | DSMB Review 2 | 10/1/2020 | 10/1/2020 | 1d | | | | | | | | | | | | | |
| 7 | DSMB Review 3 | 1/1/2021 | 1/1/2021 | 1d | | | | | | | | | | | | | |
| 8 | DSMB Review 4 | 4/1/2021 | 4/1/2021 | 1d | | | | | | | | | | | | | |

# 4) Planned data analysis

Aim 1, 2, 3: Descriptive statistics,

Compare rates of primary and secondary outcome measures in subjects receiving fluoxetine with those not receiving fluoxetine by Student t-test and Chi-square test as appropriate.

# **Data Safety Monitoring Board**

Interim data analyses will be performed every 3 months and will be presented to a 4 member data safety monitoring board who will prepare a report on the ongoing safety of the clinical trial and consideration of early termination of the study for either benefit or harm per the guidelines of Tyson et al. 2016.

#### **Reference List**

- 1. Aksu, U., Guner, I., Yaman, O. M., Erman, H., Uzun, D., Sengezer-Inceli, M., . . . Sahin, G. (2014). Fluoxetine ameliorates imbalance of redox homeostasis and inflammation in an acute kidney injury model. *J Physiol Biochem*, 70(4), 925-934. doi: 10.1007/s13105-014-0361-0
- 2. Amitai, M., Taler, M., Carmel, M., Michaelovsky, E., Eilat, T., Yablonski, M., . . . Fennig, S. (2016). The Relationship Between Plasma Cytokine Levels and Response to Selective Serotonin Reuptake Inhibitor Treatment in Children and Adolescents with Depression and/or Anxiety Disorders. *J Child Adolesc Psychopharmacol*, 26(8), 727-732. doi: 10.1089/cap.2015.0147
- 3. Bah, T. M., Benderdour, M., Kaloustian, S., Karam, R., Rousseau, G., & Godbout, R. (2011). Escitalopram reduces circulating pro-inflammatory cytokines and improves depressive behavior without affecting sleep in a rat model of post-cardiac infarct depression. *Behav Brain Res*, 225(1), 243-251. doi: 10.1016/j.bbr.2011.07.039
- 4. Baharav, E., Bar, M., Taler, M., Gil-Ad, I., Karp, L., Weinberger, A., & Weizman, A. (2012). Immunomodulatory effect of sertraline in a rat model of rheumatoid arthritis. *Neuroimmunomodulation*, 19(5), 309-318. doi: 10.1159/000339109
- 5. Basterzi, A. D., Aydemir, C., Kisa, C., Aksaray, S., Tuzer, V., Yazici, K., & Göka, E. (2005). IL-6 levels decrease with SSRI treatment in patients with major depression. *Hum Psychopharmacol*, 20(7), 473-476. doi: 10.1002/hup.717
- 6. Bertoni, S., Arcaro, V., Vivo, V., Rapalli, A., Tognolini, M., Cantoni, A. M., . . . Barocelli, E. (2014). Suppression of inflammatory events associated to intestinal ischemia-reperfusion by 5-HT1A blockade in mice. *Pharmacol Res*, 81, 17-25. doi: 10.1016/j.phrs.2014.02.002
- 7. Bhat, R., Mahapatra, S., Axtell, R. C., & Steinman, L. (2017). Amelioration of ongoing experimental autoimmune encephalomyelitis with fluoxetine. *J Neuroimmunol*, *313*, 77-81. doi: 10.1016/j.jneuroim.2017.10.012
- 8. Blatteau, J. E., Barre, S., Pascual, A., Castagna, O., Abraini, J. H., Risso, J. J., & Vallee, N. (2012). Protective effects of fluoxetine on decompression sickness in mice. *PLoS One*, *7*(11), e49069. doi: 10.1371/journal.pone.0049069
- 9. Blatteau, J. E., de Maistre, S., Lambrechts, K., Abraini, J., Risso, J. J., & Vallée, N. (2015). Fluoxetine stimulates anti-inflammatory IL-10 cytokine production and attenuates sensory deficits in a rat model of decompression sickness. *J Appl Physiol (1985), 119*(12), 1393-1399. doi: 10.1152/japplphysiol.00602.2015
- 10. Branco-de-Almeida, L. S., Kajiya, M., Cardoso, C. R., Silva, M. J., Ohta, K., Rosalen, P. L., . . Kawai, T. (2011). Selective serotonin reuptake inhibitors attenuate the antigen presentation from dendritic cells to effector T lymphocytes. *FEMS Immunol Med Microbiol*, *62*(3), 283-294. doi: 10.1111/j.1574-695X.2011.00816.x
- 11. Cai, Z., Liu, J., Bian, H., Cai, J., Jin, Q., & Han, J. (2017). Fluoxetine, an Antidepressant Drug, Inhibited Cigarette Smoke-Induced Pulmonary Inflammation and Apoptosis in Rats. *Inflammation*, 40(4), 1375-1381. doi: 10.1007/s10753-017-0580-y
- 12. Chen, C. Y., Yeh, Y. W., Kuo, S. C., Liang, C. S., Ho, P. S., Huang, C. C., . . . Huang, S. Y. (2018). Differences in immunomodulatory properties between venlafaxine and paroxetine in patients with major depressive disorder. *Psychoneuroendocrinology*, 87, 108-118. doi: 10.1016/j.psyneuen.2017.10.009
- 13. Curzytek, K., Kubera, M., Majewska-Szczepanik, M., Szczepanik, M., Marcińska, K., Ptak, W., . . . Maes, M. (2013). Inhibition of 2,4-dinitrofluorobenzene-induced contact hypersensitivity reaction by antidepressant drugs. *Pharmacol Rep*, 65(5), 1237-1246. doi: 10.1016/s1734-1140(13)71481-6
- 14. Dong, C., Zhang, J. C., Yao, W., Ren, Q., Yang, C., Ma, M., . . . Hashimoto, K. (2016). Effects of escitalopram, R-citalopram, and reboxetine on serum levels of tumor necrosis factor-α,

- interleukin-10, and depression-like behavior in mice after lipopolysaccharide administration. *Pharmacol Biochem Behav, 144*, 7-12. doi: 10.1016/j.pbb.2016.02.005
- 15. Durairaj, H., Steury, M. D., & Parameswaran, N. (2015). Paroxetine differentially modulates LPS-induced TNFα and IL-6 production in mouse macrophages. *Int Immunopharmacol*, *25*(2), 485-492. doi: 10.1016/j.intimp.2015.02.029
- 16. Ehret, M., & Sobieraj, D. M. (2014). Prevention of interferon-alpha-associated depression with antidepressant medications in patients with hepatitis C virus: a systematic review and meta-analysis. *Int J Clin Pract*, 68(2), 255-261. doi: 10.1111/jjcp.12268
- 17. Gałecki, P., Mossakowska-Wójcik, J., & Talarowska, M. (2018). The anti-inflammatory mechanism of antidepressants SSRIs, SNRIs. *Prog Neuropsychopharmacol Biol Psychiatry*, 80(Pt C), 291-294. doi: 10.1016/j.pnpbp.2017.03.016
- 18. Gobin, V., Van Steendam, K., Denys, D., & Deforce, D. (2014). Selective serotonin reuptake inhibitors as a novel class of immunosuppressants. *Int Immunopharmacol*, 20(1), 148-156. doi: 10.1016/j.intimp.2014.02.030
- 19. Hashioka, S., Klegeris, A., Monji, A., Kato, T., Sawada, M., McGeer, P. L., & Kanba, S. (2007). Antidepressants inhibit interferon-gamma-induced microglial production of IL-6 and nitric oxide. *Exp Neurol*, 206(1), 33-42. doi: 10.1016/j.expneurol.2007.03.022
- 20. Horikawa, H., Kato, T. A., Mizoguchi, Y., Monji, A., Seki, Y., Ohkuri, T., . . . Kanba, S. (2010). Inhibitory effects of SSRIs on IFN-γ induced microglial activation through the regulation of intracellular calcium. *Prog Neuropsychopharmacol Biol Psychiatry*, *34*(7), 1306-1316. doi: 10.1016/j.pnpbp.2010.07.015
- 21. Hu, T. M., Subeq, Y. M., Yang, F. L., Hsu, B. G., Lin, N. T., & Lee, R. P. (2013). The use of a selective serotonin reuptake inhibitor decreases heavy alcohol exposure-induced inflammatory response and tissue damage in rats. *J Psychopharmacol*, *27*(10), 940-946. doi: 10.1177/0269881113494938
- 22. Koh, S. J., Kim, J. M., Kim, I. K., Kim, N., Jung, H. C., Song, I. S., & Kim, J. S. (2011). Fluoxetine inhibits NF-κB signaling in intestinal epithelial cells and ameliorates experimental colitis and colitis-associated colon cancer in mice. *Am J Physiol Gastrointest Liver Physiol*, *301*(1), G9-19. doi: 10.1152/ajpgi.00267.2010
- 23. Koh, S. J., Kim, J. W., Kim, B. G., Lee, K. L., Im, J. P., & Kim, J. S. (2015). Fluoxetine inhibits hyperresponsive lamina propria mononuclear cells and bone marrow-derived dendritic cells, and ameliorates chronic colitis in IL-10-deficient mice. *Dig Dis Sci, 60*(1), 101-108. doi: 10.1007/s10620-014-3326-9
- 24. Kubera, M., Kenis, G., Bosmans, E., Kajta, M., Basta-Kaim, A., Scharpe, S., . . . Maes, M. (2004). Stimulatory effect of antidepressants on the production of IL-6. *Int Immunopharmacol*, *4*(2), 185-192. doi: 10.1016/j.intimp.2003.11.006
- 25. Li, X. Q., Wang, H. M., Yang, C. G., Zhang, X. H., Han, D. D., & Wang, H. L. (2011). Fluoxetine inhibited extracellular matrix of pulmonary artery and inflammation of lungs in monocrotaline-treated rats. *Acta Pharmacol Sin*, 32(2), 217-222. doi: 10.1038/aps.2010.187
- 26. Liechti, F. D., Grandgirard, D., & Leib, S. L. (2015). The antidepressant fluoxetine protects the hippocampus from brain damage in experimental pneumococcal meningitis. *Neuroscience*, 297, 89-94. doi: 10.1016/j.neuroscience.2015.03.056
- 27. Liu, D., Wang, Z., Liu, S., Wang, F., Zhao, S., & Hao, A. (2011). Anti-inflammatory effects of fluoxetine in lipopolysaccharide(LPS)-stimulated microglial cells. *Neuropharmacology*, *61*(4), 592-599. doi: 10.1016/j.neuropharm.2011.04.033
- 28. Liu, F. Y., Cai, J., Wang, C., Ruan, W., Guan, G. P., Pan, H. Z., . . . Chen, G. (2018). Fluoxetine attenuates neuroinflammation in early brain injury after subarachnoid hemorrhage: a possible role for the regulation of TLR4/MyD88/NF-κB signaling pathway. *J Neuroinflammation*, *15*(1), 347. doi: 10.1186/s12974-018-1388-x

- 29. Liu, R. P., Zou, M., Wang, J. Y., Zhu, J. J., Lai, J. M., Zhou, L. L., . . . Zhu, J. H. (2014). Paroxetine ameliorates lipopolysaccharide-induced microglia activation via differential regulation of MAPK signaling. *J Neuroinflammation*, 11, 47. doi: 10.1186/1742-2094-11-47
- 30. Lu, Y., Xu, X., Jiang, T., Jin, L., Zhao, X. D., Cheng, J. H., . . . Piao, L. X. (2019). Sertraline ameliorates inflammation in CUMS mice and inhibits TNF-α-induced inflammation in microglia cells. *Int Immunopharmacol*, *67*, 119-128. doi: 10.1016/j.intimp.2018.12.011
- 31. Pizzi, C., Mancini, S., Angeloni, L., Fontana, F., Manzoli, L., & Costa, G. M. (2009). Effects of selective serotonin reuptake inhibitor therapy on endothelial function and inflammatory markers in patients with coronary heart disease. *Clin Pharmacol Ther*, 86(5), 527-532. doi: 10.1038/clpt.2009.121
- 32. Roumestan, C., Michel, A., Bichon, F., Portet, K., Detoc, M., Henriquet, C., . . . Mathieu, M. (2007). Anti-inflammatory properties of desipramine and fluoxetine. *Respir Res*, *8*, 35. doi: 10.1186/1465-9921-8-35
- 33. Sacre, S., Medghalchi, M., Gregory, B., Brennan, F., & Williams, R. (2010). Fluoxetine and citalopram exhibit potent antiinflammatory activity in human and murine models of rheumatoid arthritis and inhibit toll-like receptors. *Arthritis Rheum*, 62(3), 683-693. doi: 10.1002/art.27304
- 34. Sherkawy, M. M., Abo-Youssef, A. M., Salama, A. A. A., & Ismaiel, I. E. (2018). Fluoxetine protects against OVA induced bronchial asthma and depression in rats. *Eur J Pharmacol*, 837, 25-32. doi: 10.1016/j.ejphar.2018.08.026
- 35. Taler, M., Gil-Ad, I., Korob, I., & Weizman, A. (2011). The immunomodulatory effect of the antidepressant sertraline in an experimental autoimmune encephalomyelitis mouse model of multiple sclerosis. *Neuroimmunomodulation*, 18(2), 117-122. doi: 10.1159/000321634
- 36. Taraz, M., Khatami, M. R., Dashti-Khavidaki, S., Akhonzadeh, S., Noorbala, A. A., Ghaeli, P., & Taraz, S. (2013). Sertraline decreases serum level of interleukin-6 (IL-6) in hemodialysis patients with depression: results of a randomized double-blind, placebo-controlled clinical trial. *Int Immunopharmacol*, 17(3), 917-923. doi: 10.1016/j.intimp.2013.09.020
- 37. Tousoulis, D., Drolias, A., Antoniades, C., Vasiliadou, C., Marinou, K., Latsios, G., . . . Stefanadis, C. (2009). Antidepressive treatment as a modulator of inflammatory process in patients with heart failure: effects on proinflammatory cytokines and acute phase protein levels. *Int J Cardiol*, 134(2), 238-243. doi: 10.1016/j.ijcard.2008.02.013
- 38. Tsai, J. H., Kuo, C. H., Yang, P., Cheng, K. H., Wang, P. W., Chen, C. C., & Hung, C. H. (2014). Effects of antidepressants on IP-10 production in LPS-activated THP-1 human monocytes. *Int J Mol Sci*, *15*(8), 13223-13235. doi: 10.3390/ijms150813223
- 39. Tynan, R. J., Weidenhofer, J., Hinwood, M., Cairns, M. J., Day, T. A., & Walker, F. R. (2012). A comparative examination of the anti-inflammatory effects of SSRI and SNRI antidepressants on LPS stimulated microglia. *Brain Behav Immun*, 26(3), 469-479. doi: 10.1016/j.bbi.2011.12.011
- 40. Udina, M., Hidalgo, D., Navinés, R., Forns, X., Solà, R., Farré, M., . . . Martín-Santos, R. (2014). Prophylactic antidepressant treatment of interferon-induced depression in chronic hepatitis C: a systematic review and meta-analysis. *J Clin Psychiatry*, 75(10), e1113-1121. doi: 10.4088/JCP.13r08800
- 41. Uher, R., Perroud, N., Ng, M. Y., Hauser, J., Henigsberg, N., Maier, W., . . . McGuffin, P. (2010). Genome-wide pharmacogenetics of antidepressant response in the GENDEP project. *Am J Psychiatry*, 167(5), 555-564. doi: 10.1176/appi.ajp.2009.09070932
- 42. van Noort, V., Schölch, S., Iskar, M., Zeller, G., Ostertag, K., Schweitzer, C., . . . Bork, P. (2014). Novel drug candidates for the treatment of metastatic colorectal cancer through global inverse gene-expression profiling. *Cancer Res*, 74(20), 5690-5699. doi: 10.1158/0008-5472.CAN-13-3540
- 43. Vollmar, P., Haghikia, A., Dermietzel, R., & Faustmann, P. M. (2008). Venlafaxine exhibits an anti-inflammatory effect in an inflammatory co-culture model. *Int J Neuropsychopharmacol*, 11(1), 111-117. doi: 10.1017/S1461145707007729

- 44. Wang, L., Wang, R., Liu, L., Qiao, D., Baldwin, D. S., & Hou, R. (2019). Effects of SSRIs on peripheral inflammatory markers in patients with major depressive disorder: A systematic review and meta-analysis. *Brain Behav Immun*, 79, 24-38. doi: 10.1016/j.bbi.2019.02.021
- 45. Wang, Y., Gu, Y. H., Liu, M., Bai, Y., & Wang, H. L. (2017). Fluoxetine protects against methamphetamine-induced lung inflammation by suppressing oxidative stress through the SERT/p38 MAPK/Nrf2 pathway in rats. *Mol Med Rep, 15*(2), 673-680. doi: 10.3892/mmr.2016.6072
- 46. Więdłocha, M., Marcinowicz, P., Krupa, R., Janoska-Jaździk, M., Janus, M., Dębowska, W., . . Szulc, A. (2018). Effect of antidepressant treatment on peripheral inflammation markers A meta-analysis. *Prog Neuropsychopharmacol Biol Psychiatry*, 80(Pt C), 217-226. doi: 10.1016/j.pnpbp.2017.04.026
- 47. Young, K. C., Bai, C. H., Su, H. C., Tsai, P. J., Pu, C. Y., Liao, C. S., . . . Tsao, C. W. (2014). Fluoxetine a novel anti-hepatitis C virus agent via ROS-, JNK-, and PPARβ/γ-dependent pathways. *Antiviral Res*, *110*, 158-167. doi: 10.1016/j.antiviral.2014.08.002
- 48. Yuan, X. Q., Qiu, G., Liu, X. J., Liu, S., Wu, Y., Wang, X., & Lu, T. (2012). Fluoxetine promotes remission in acute experimental autoimmune encephalomyelitis in rats. *Neuroimmunomodulation*, 19(4), 201-208. doi: 10.1159/000334095